CLINICAL TRIAL: NCT03552848
Title: Mesenchymal Stem Cells for Multiple Organ Dysfuntion Syndrome After Surgical Repaire of Acute Type A Aortic Dissection: a Pilot Study
Brief Title: Mesenchymal Stem Cells for Multiple Organ Dysfuntion Syndrome After Surgical Repaire of Acute Type A Aortic Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Liang-Wan Chen MD, Department Director, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018005
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Multiple Organ Dysfunction Syndrome
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Intervention Model Description: Part 1: totally 30 patient will be enrolled, and 15 patients will be given MSC immediately after ascending aortic replacement combined with open placement of triple-branched stent graft for ATAAD.
  Part 2: totally 30 patient will be enrolled, and 15 patients will be given MSC after onset of multiple organ dysfuntion syndrome after ascending aortic replacement combined with open placement of triple-branched stent graft for ATAAD.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cell (Experimental): Patients in the MSC arm will be given MSC, i.v., 1000000 cells per kilogram of body weight.
  Interventions: Biological: MSC
- Control (No Intervention): Patients in the control arm will not be given MSC.

INTERVENTIONS:
Biological: MSC — MSC at a dose of 1000000 cells per kilogram of body weight will be given intravenously once every 4 days for 4 times
  Arms: Mesenchymal stem cell

SUMMARY:
Multiple organ dysfunction syndrome (MODS) after surgical repaire for acute type A aortic dissection(ATAAD) is a life-threatening condition. In this study, patients who undergoing surgical repaire of ATAAD immdediately or presenting sever MODS after surgical repaire of acute type A aortic dissection will be treated with umbilical cord-derived mesenchymal stem cell.

DETAILED DESCRIPTION:
Multiple organ dysfunction syndrome(MODS) are common debilitating complications after surgical repaire for ATAAD. MODS is one of the chief causes of post-operative death for acute type A aortic dissection(ATAAD) patients, and it was reported that MODS accounted for more than half of the death after surgery for ATAAD. Despite recent advance in surgical technique, mortality rate remains high in such critical care conditions.

In animal models, studies have demonstrated the beneficial effects of MSCs with respect to ischemia-reperfusion injury of heart, lungs, kidney, brains and livers. Several pilot studies have provided evidence that MSC may be effective in treating critically ill patients with traumatic brain injury, acute renal failure, or acute respiratory distress syndrome. Therefore, in the present pilot study, the investigators hypothesized that timely initiation of mesenchymal stem cells(MSC) will positively influence survival and biochemical indexesof patients with MODS after ascending aortic replacement combined with open placement of triple-branched stent graft for ATAAD. The trial contain two parts:

Part one(prenvention scheme): to explore the safety and efficacy of umbilical cord-derived MSC, we will recruit patients who are diagnosed with ATAAD, and 8 patients will be administrated intervenously with MSC immediately after ascending aortic replacement combined with open placement of triple-branched stent graft while other 8 not. Then we will monitor their MODS related biochemical indexes, sequential organ failure assessment(SOFA) scores, comparing to those don't be treated with MSC.

Phase two(treatment scheme): for patients presenting severe MODS(SOFA score≥10) after ascending aortic replacement combined with open placement of triple-branched stent graft, we will randomly use MSC to 8 of patients while other 8 not. Then we will monitor their MODS related biochemical indexes, SOFA scores, comparing to those don't be treated with MSC.

The dosage of the MSC was determined on the basis of the previous clinical studies, which is 1000000 cells per kilogram of body weight and administrated intervenously .

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Patients who are diagnosed with ATAAD and received emergency surgery with ascending aortic replacement combined with open placement of triple-branched stent graft
* elder than 60 years old
* Preoperative PaO2/FiO2 > 400mmHg, platelets ≥ 150*109/L, bilirubin < 20μmol/L, no hypotension (without vasoactive drugs), Glasgow Coma Score Scale = 15, creatine <110μmol/L

Part 2:

* Patients who are diagnosed with ATAAD and received emergency surgery with ascending aortic replacement combined with open placement of triple-branched stent graft
* Patients who have failure of at least 2 organs
* Patients who meet the criteria as below:

sequential organ failure assessment score (SOFA) ≥ 10

Exclusion Criteria:

* uncontrollable underlying disease life expectancy of less than 4 days history of long-term corticosteroid use during the past 6 months.
* The pre-operative computer tomography angiography(CTA) demonstrate the visceral arteries are involved
* pre-existing severe disease of any major organs

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
survival after intervention | Up to 6 month
  survival after intervention: comparing survival ratio in hospital(6 months post-intervention) between groups.
adverse events | Up to 2 years
  short term adverse events such as anaphylactic reaction, embolism; long term adverse events, such as oncogenicity
sequential organ failure assessment score(SOFA) | Up to 6 months
  Compare the change of sequential organ failure assessment score(SOFA) between groups.
interleukin-6 | Early 3 days
  Compare the change of interleukin( IL)-6 between groups.

SECONDARY OUTCOMES:
the effects on kidney function | Up to 6 months
  the therapeutic effects in the improvement of kidney function, as indicated by Scr level.
the effects on liver function | Up to 6 months
  the therapeutic effects in the improvement of liver function, as indicated by bilirubin levels.
the effects on lung function | Up to 6 months
  the therapeutic effects in the improvement of lung function, as indicated by oxygenation index.
the effects on coagulation function | Up to 6 months
  the therapeutic effects in the improvement of coagulation function, as indicated by blood platelet count.
the effects on central nervous system | Up to 6 months
  the therapeutic effects in the improvement of coagulation function, as indicated by Glosgow coma score

CONTACTS AND LOCATIONS:
Overall Officials: Liangwan Chen, M.D, Principal Investigator — Union Hospital
Locations (1):
- Department of Cardiovascular Surgery, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No